CLINICAL TRIAL: NCT02177656
Title: Motivational Interviewing Tailored Intervention for Patients With Heart Failure (MITI-HF)
Acronym: MITI-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruth Masterson-Creber (Other)
Collaborators: Edna G Kynett Memorial Foundation (Unknown); University of Pennsylvania (Other)
Responsible Party: Sponsor-Investigator, Ruth Masterson-Creber, Pre-doctoral student in Nursing Science at the University of Pennsylvania, University of Pennsylvania
Organization: University of Pennsylvania (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MITI-HF_EGKMF
Record Dates: First submitted 2014-06-13; First posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
Keywords: heart failure; self-care; self-care maintenance; self-care management; self-efficacy; quality of life; symptoms
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (No Intervention): Patients in the usual care group received six patient educational materials in the hospital, a baseline and follow-up phone call by blinded research assistants.
- MI tailored intervention (Experimental): The MI intervention was provided by a heart failure specialist nurse. The nurse conducted a home-based motivational interviewing intervention followed up by three phone calls over the course of 90 days. The intervention began with a conversation about the participant's self-identified goals. In the home intervention, the nurse focused on self-care areas that the participant identified as high priority. During the home-based intervention, the participant also set specific goals, which the nurse followed up with and reinforced over the follow-up phone calls.
  Interventions: Behavioral: Motivational Interviewing tailored intervention

INTERVENTIONS:
Behavioral: Motivational Interviewing tailored intervention — MI is grounded in client-centered counseling, cognitive-behavioral therapy, and social cognitive therapy. MI integrates the concepts of relationship building from humanistic therapy with active strategies oriented towards stages of change.The main characteristics of motivational interviewing are: expressing empathy, developing discrepancy, rolling with resistance, and supporting self-efficacy. The interviewer maintains a nonjudgmental approach and allows the patient to determine the need for behavioral change, rather than offering unsolicited advice on the need for change. The interviewer only explores ways to implement change once the patient expresses the desire and confidence to change. The goal of MI is to help individuals work through inherent ambivalence present in problematic or unhealthy behaviors and to help them verbally express reasons for or against change using a nonjudgmental, empathetic and encouraging tone.
  Arms: MI tailored intervention

SUMMARY:
This study will test the effectiveness of motivational interviewing and skill building compared to usual care to improve self-care in heart failure (HF) patients. The target population is HF patients recruited from the Hospital of the University of Pennsylvania after an in-patient admission. Patients in the intervention arms will receive one home-visit from a nurse who does a self-care intervention followed up by 3 follow-up phone calls.

DETAILED DESCRIPTION:
MITI-HF is a prospective, single blinded, pilot randomized single-site trial. The target sample size was 65 participants; however, to account for an estimated 35% attrition rate, the target number for recruitment was 100 participants. We calculated the target sample size based on a 2:1 randomization (intervention: control) with 90% power (5% alpha) to detect a difference of 80% versus 50% (intervention and control group) of scoring over 70, which is the cut-off for adequate self-care at three months between the two groups. The power analysis was performed using G*Power and confirmed with PASS. Randomization to the intervention or usual care group occurred after the informed consent form was signed and New York Heart Association (NYHA) Functional Class was scored. To achieve balance in both arms of the study, the Minim randomization program was used to minimize prognostic factor differences between groups. Minim stratified participants based on NYHA class and gender to one of two arms in a 2:1 ratio (intervention: control). The research assistants were blinded to group assignment until all study data was collected. All eligible patients were screened for health literacy using a three-question health literacy questionnaire, cognitive impairment using a six-item screener derived from the Mini Mental Status Exam (MMSE), baseline self-care using the SCHFI (v.6.2), and NYHA functional class using the Central Assessment of NYHA Functional Class. A single board-certified cardiologist scored all of the NYHA functional class scores. Medical, socio-demographic, Kansas City Cardiomyopathy Questionnaire (KCCQ), and Heart Failure Somatic Perception Scale (HFSPS) data were collected at baseline via phone call by blinded research assistants (RA) approximately two weeks after hospital discharge. Socio-demographics were assessed using a questionnaire that inquires about gender, age, marital/partnership status, ethnicity/race, and employment. Follow-up data were collected at 90 days by the blinded RAs. If the first call was unsuccessful, the RA would try every 3 to 5 days for up to 60 days. If there was no contact with the participant after 60 days from the expected follow-up date, the participant was considered lost to follow-up. During the follow-up phone call, participants completed the SCHFI, KCCQ, HFSPS and self-reported clinical events within the study period. Self-reported clinical events were verified with a review of the electronic medical record to confirm any hospitalizations, emergency room visits, or outpatient heart failure related visits that occurred within the study period.

ELIGIBILITY:
Inclusion Criteria:

To be included, participants had to be:

1. hospitalized with a primary or secondary diagnosis of heart failure
2. able to read and speak English
3. 18 years of age or older
4. living in a setting where they can independently engage in self-care
5. living within 30 miles from the University hospital
6. have at least adequate health literacy
7. symptomatic HF (NYHA II-IV)
8. willing to participate

Exclusion Criteria:

Exclusion criteria included:

1. being on a Milrinone drip
2. being on a list for an implanted ventricular assist device or heart transplant
3. pregnancy
4. psychosis
5. cognitive impairment with the inability to participate in the intervention or complete the study instruments
6. inability to provide informed consent

Study enrollment took place from January 2012 to December 2013.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
self-care maintenance | baseline, 90 days
  Self-Care will be self-reported and measured using the Self-Care of Heart Failure Index (SCHFI). Items measuring self-care maintenance address treatment adherence and self-monitoring, while management focuses on decision-making in response to symptoms. Higher scores reflect better self-care maintenance. Each scale is scored separately; the total possible score for each scale is 100.
self-care management | baseline, 90 days
  Self-Care management will be self-reported and measured using the Self-Care of Heart Failure Index (SCHFI). Self care management is a patients ability to recognize symptoms when they occur; independent and interdependent self-care treatments implemented by the patient (e.g., take an extra diuretic for shortness of breath) and ability to evaluate the effectiveness of the treatments implemented. Higher scores reflect better self-care. Each scale is scored separately; the total possible score for each scale is 100.
self-care confidence | baseline, 90 days
  Self-Care confidence will be self-reported and measured using the Self-Care of Heart Failure Index (SCHFI). The SCHFI captures confidence in the ability to perform self-care.

SECONDARY OUTCOMES:
Quality of life | baseline and 90 days
  Quality of Life will be measured with the Kansas City Cardiomyopathy Questionnaire (KCCQ), a 23-item questionnaire that quantifies disease-specific physical limitation, symptom frequency, severity, and change over time, overall quality of life, social interference, and self-efficacy and knowledge.
Somatic symptom awareness | baseline and 90 days
  Somatic Awareness will be measured using the 18-item HF Somatic Perception Scale (HFSAS).
Hospitalizations | baseline and 90 days
  Hospitalizations were self-reported at 90 days and verified with the medical record.

CONTACTS AND LOCATIONS:
Overall Officials: Ruth M Masterson Creber, MSc RN PhD (c), Principal Investigator — University of Pennsylvania; Barbara Riegel, DNSc, RN, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States